CLINICAL TRIAL: NCT06425913
Title: Short-Term Effects of Cold Therapy and Kinesio Taping on Pain and Upper Extremity Functionality in Individuals With Rotator Cuff Tendonitis: A Randomized Study
Brief Title: Effects of Cold and Kinesio Taping in Individuals With Rotator Cuff Tendonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Elif Durgut, Asst. Prof, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71306642
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Rotator Cuff Tendinitis
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants were unaware of their group assignments. A therapist who was unaware of the intervention protocol and assigned groups performed the assessment procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (Active Comparator): KT was applied to the symptomatic shoulder of participants.
  Interventions: Other: Kinesio Taping (KT); Other: standardized home exercise program
- Cold Therapy (Active Comparator): Ice packs were applied to the symptomatic shoulder of participants.
  Interventions: Other: Cold Therapy (CT); Other: standardized home exercise program

INTERVENTIONS:
Other: Kinesio Taping (KT) — KT was applied to the symptomatic shoulder at the end of the baseline assessment by a certificated physiotherapist with over ten years of experience in Kinesio taping. After three days, participants were re-evaluated. KT application has been made according to the protocol for rotator cuff impingement or tendonitis including inhibition and correction techniques.
  Arms: Kinesio Taping
Other: Cold Therapy (CT) — The initial application was administered by the physiotherapist. In a sitting position, a pack was wrapped in a thin towel and placed on the affected shoulder joint, including the painful locations. During the application, the participant was closely observed for discomfort or adverse reactions (redness, burning, numbness, itching, …). The cold application was continued for 20 minutes.After the first application, participants were instructed to apply ice for 20 minutes five times a day for three days at home or work.
  Arms: Cold Therapy
Other: standardized home exercise program — All participants performed standardized home exercise program, including shoulder isometric and stretching exercises were . A physiotherapist taught the exercise program until the participants were able to exercise accurately on their own. All participants were instructed to perform the exercises three times a day for three days.

SUMMARY:
Rotator cuff tendonitis (RCT) is one of the most common shoulder pathologies, causing pain, limitation of shoulder joint movements, and impaired function. Patient education, medical treatment, corticosteroid injections, physiotherapy rehabilitation approaches are the most common treatment options applied to alleviate the symptoms of RCT. Despite these various treatment methods, there are currently no specific guidelines regarding the most appropriate and effective intervention for RCT treatment. This is mainly because adequate, high-quality studies are lacking in RCT management. To the best of our knowledge, no studies have evaluated the effects of Kinesio Taping (KT), which has become a popular approach in recent years, and Cold Therapy (CT), which has often been used as a therapeutic agent since immemorial, on individuals with RCT. In this regard, this study aimed to investigate and compare the short-term effects of KT and CT on pain and upper extremity functionality in individuals with RCT.

ELIGIBILITY:
Inclusion Criteria:

* RCT diagnosis
* Excluding other shoulder pathologies by magnetic resonance imaging (MRI) and specific tests

Exclusion Criteria:

* Glenohumeral joint dislocation/subluxation;
* Acromioclavicular sprain;
* Rotator cuff tear;
* Glenohumeral joint instability;
* Calcific tendinitis of the shoulder;
* Acromioclavicular joint pathologies,
* Hyperlaxity;
* Any fracture in the shoulder;
* Diabetes, thyroid and any vascular or rheumatologic disease;
* Glenohumeral joint deformities;
* Superior labrum anteroposterior (SLAP) lesion;
* Shoulder pain lasting more than six months;
* History of shoulder surgery;
* Intra-articular steroid injection

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | At baseline and after three days of the applications
  Numerical Rating Scale (NRS): The pain severity was assessed using the NRS, for which a subject was asked to rate his/her perceived pain. A 11-point NRS from 0 to 10 which 0 means no pain and 10 means the worst possible pain was scored during night, rest, and activity.
Function | At baseline and after three days of the applications
  Disability of the Arm, Shoulder and Hand (DASH) Questionnaire): DASH is a self-reported questionnaire designed for evaluating the functional level of upper extremity. It is a 30-item scale that addresses difficulty in performing various physical activities that require upper extremity function (physical function, 21 items); symptoms of pain, activity-related pain, tingling, weakness, and stiffness (pain symptoms, 5 items); or impact of disability and symptoms on social activities, work, sleep, and psychological well-being (emotional and social function, 4 items). Each item is scored between 1 and 5. A score of 1 indicates no strain, and a score of 5 indicates inability to perform the specified activity.
Function | At baseline and after three days of the applications
  Shoulder Pain and Disability Index (SPADI): The SPADI is a self-administered questionnaire developed to measure the pain and disability associated with shoulder pathology in people with shoulder pain of musculoskeletal, neurogenic, or undetermined origin. It consists of 13 items that assess two domains: a 5-item subscale that measures pain and an 8-item subscale that measures disability. The items of both domains were scored on a numerical rating scale ranging from 0 to 10, where 0=no pain/no disability and 10= worst pain imaginable/so difficult required help.

SECONDARY OUTCOMES:
Range of Motion | At baseline and after three days of the applications
  Range of Motion (ROM): The active range of motion (ROM) of the affected shoulder, including flexion, abduction, external rotation, and internal rotation, was assessed using a universal goniometer following the protocol reported by the American Academy of Orthopaedic Surgeons (AAOS)
Grip strength | At baseline and after three days of the applications
  Jamar® hydraulic hand dynamometer were used to assess hand-grip strength of the affected side.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared